CLINICAL TRIAL: NCT03896945
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-arm Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Negative Symptoms of Schizophrenia
Brief Title: Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Negative Symptoms of Schizophrenia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Based on the Interim Analysis outcome and recommendation by the DMC, Otsuka approved termination of the study based on futility.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-AVP-786-207; 2021-001352-33 (EudraCT Number)
Record Dates: First submitted 2019-03-19; First posted 2019-04-01 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia
Keywords: Negative Symptoms; Schizophrenia; AVP-786
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules will be administered orally twice a day over a 15-week period.
  Interventions: Drug: Placebo
- AVP-786 (Experimental): AVP-786 capsules will be administered orally twice a day over a 15-week period.
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: Placebo — oral capsules
  Arms: Placebo
Drug: AVP-786 — oral capsules
  Arms: AVP-786

SUMMARY:
This study will be conducted to evaluate the efficacy, safety, and tolerability of AVP-786, as compared with placebo, for the treatment of negative symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) diagnostic criteria for schizophrenia confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I) Version 7.0.2
* Participants must have well-controlled positive symptoms and prominent negative symptoms as defined by Positive and Negative Syndrome Scale (PANSS) criteria.
* Participants currently receiving a second-generation atypical antipsychotic drug (SGA) are eligible if they are stable and adherent to their dosing schedule.
* Participants must have a reliable informant (e.g., case manager, social worker, family member). The informant should be able to spend an adequate amount of time with the participant to be able to address behaviors, activities, and symptoms.

Exclusion Criteria:

* Participants with current major depressive disorder (MDD)
* Participants with pseudo-parkinsonism secondary to their ongoing antipsychotic medication
* Participants currently using anticholinergic medications
* Participants recently hospitalized as in-patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 15 in the Positive and Negative Syndrome Scale (PANSS) Marder Negative Factors Score | Baseline; Week 15

SECONDARY OUTCOMES:
Change from Baseline to Week 15 in the Negative Symptom Assessment-16 (NSA-16) Global Negative Symptom Score | Baseline; Week 15
Change from Baseline to Week 15 in the Patient Global Impression of Severity (PGI-S) Score | Baseline; Week 15
Change from Baseline to Week 15 in the Patient Global Impression of Change (PGI-C) Score | Baseline; Week 15

CONTACTS AND LOCATIONS:
Locations (72):
- United States (61):
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site #840-041, Anaheim, California
  - Clinical Research Site #840-013, Bellflower, California
  - Clinical Research Site #840-079, Costa Mesa, California
  - Clinical Research Site #840-027, Culver City, California
  - Clinical Research Site #840-006, Garden Grove, California
  - Clinical Research Site #840-026, Glendale, California
  - Clinical Research Site# 840-067, La Habra, California
  - Clinical Research Site# 840-083, Lafayette, California
  - Clinical Research Site 840-002, Lemon Grove, California
  - Clinical Research Site, Oakland, California
  - Clinical Research Site #840-035, Oceanside, California
  - Clinical Research Site# 840-010, Panorama City, California
  - Clinical Research Site #840-012, Riverside, California
  - Clinical Research Site# 840-081, San Bernardino, California
  - Clinical Research Site #840-005, San Diego, California
  - Clinical Research Site #840-096, Santee, California
  - Clinical Research Site #840-015, Torrance, California
  - Clinical Research Site# 840-094, Doral, Florida
  - Clinical Research Site #840-046, Hollywood, Florida
  - Clinical Research Site Site #840-093, Homestead, Florida
  - Clinical Research Site #840-062, Lakeland, Florida
  - Clinical Research Site #840-024, Largo, Florida
  - Clinical Research Site #840-032, Miami, Florida
  - Clinical Research Site #840-080, Miami, Florida
  - Clinical Research Site #840-084, Miami Lakes, Florida
  - Clinical Research Site, Okeechobee, Florida
  - Clinical Research Site # 840-102, Weston, Florida
  - Clinical Research Site #840-088, Atlanta, Georgia
  - Clinical Research Site #840-091, Atlanta, Georgia
  - Clinical Research Site #840-008, Atlanta, Georgia
  - Clinical Research Site #840-063, Decatur, Georgia
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site #840-090, Springfield, Illinois
  - Clinical Research Site, Lake Charles, Louisiana
  - Clinical Research Site #840-098, Shreveport, Louisiana
  - Clinical Research Site #840-072, Worcester, Massachusetts
  - Clinical Research Site #840-057, Flowood, Mississippi
  - Clinical Research Site #840-040, Olivette, Missouri
  - Clinical Research Site #840-029, Saint Charles, Missouri
  - Clinical Research Site #840-034, Saint Charles, Missouri
  - Clinical Research Site, St Louis, Missouri
  - Clinical Research Site #840-025, St Louis, Missouri
  - Clinical Research Site #840-028, Berlin, New Jersey
  - Clinical Research Site #840-009, Jamaica, New York
  - Clinical Research Site #840-070, New York, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site #840-074, Charlotte, North Carolina
  - Clinical Research Site #840-052, Middleburg Heights, Ohio
  - Clinical Research Site, Edmond, Oklahoma
  - Clinical Research Site #840-065, Oklahoma City, Oklahoma
  - Clinical Research Site #840-061, Media, Pennsylvania
  - Clinical Research Site, Norristown, Pennsylvania
  - Clinical Research Site #840-099, Myrtle Beach, South Carolina
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, DeSoto, Texas
  - Clinical Research Site #840-058, Fort Worth, Texas
  - Clinical Research Site #840-018, Richardson, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site #840-069, Springville, Utah
  - Clinical Research Site #840-051, Everett, Washington
- Bulgaria (6):
  - Clinical Research Site #009, Kazanlak
  - Clinical Research Site #100-008, Novi Iskar
  - Clinical Research Site #100-007, Plovdiv
  - Clinical Research Site #100-004 2, Sofia
  - Clinical Research Site #100-006, Veliko Tarnovo
  - Clinical Research Site #100-001, Vratsa
- Poland (3):
  - Clinical Research Site, Tuszyn, Woj.Iodzkie
  - Clinical Research Site #616-002, Bełchatów
  - Clinical Research Site #616-003, Pruszcz Gdański
- Puerto Rico (2):
  - Clinical Research Site #630-001, San Juan
  - Clinical Research Site # 630-002, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com